CLINICAL TRIAL: NCT00496743
Title: A Prospective, Open-Label Study on Low-Dose Total Skin Electron Beam Therapy in Mycosis Fungoides
Brief Title: Study of Low-Dose Total Skin Electron Beam Therapy in Mycosis Fungoides
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was discontinued after the first 10 patients because of discouraging results.
Sponsor: Bispebjerg Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-235/01
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Last update posted 2007-07-04 (Estimated); Status verified 2007-07

CONDITIONS: Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Low-dose total skin electron beam therapy (4 Gy)

SUMMARY:
The purpise of this study was to determine the effect of low-dose (4 Gy) total skin electron beam therapy as a second-line treatment of stage IB-II mycosis fungoides.

DETAILED DESCRIPTION:
Current treatment modalities are usually not curative and having treatment options suitable for the long-term control therefore essential. Electron beam therapy is generally applied to the skin in total doses of 30-36 Gy over a 8-10 week period.Due to the potential risk of toxicity including bone marrow supression, no more than 2-3 courses in a life time are generally recommended. In the current study we explored the possibility of using lower radiation doses for total skin electron beam therapy for long-term disease control.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed mycosis fungoides stage I-II with failure to obtain full remission after standard PUVA treatment or relapse within 4 months of PUVA treatment

Exclusion Criteria:

* under 18 years, pregnancy, other somatic diseases with a life expentancy under 1/2 years, psycological disorder preventing the patient to understand the information and cooperate in the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-01; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Response rates
Duration of responses

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gniadecki, MD, Principal Investigator — Bispebjerg Hospital